CLINICAL TRIAL: NCT05600335
Title: Short-term Outcomes of Enhanced Recovery After Surgery Protocol in Robotic-assisted McKeown Esophagectomy for Esophageal Cancer
Brief Title: Short-term Outcomes of ERAS Protocol in RAME for Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiajun Xiong, MD, West China Hospital
Other Study IDs: HXDB-1908
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Cancer Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS group
  Interventions: Procedure: ERAS protocol
- Conventional group
  Interventions: Procedure: ERAS protocol

INTERVENTIONS:
Procedure: ERAS protocol — Patients with esophageal cancer have undergone RAME using ERAS protocol and conventional management strategy

SUMMARY:
This single-center, retrospective cohort study aimed to evaluate the short-term outcomes of enhanced recovery after surgery (ERAS) protocol in perioperative robotic-assisted McKeown esophagectomy (RAME) among esophageal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. first detected and endoscopically confirmed esophageal cancer;
2. preoperative evaluation showed no distant metastases and suitable for RAME;
3. preoperative clinical stage of I to III;

Exclusion Criteria:

1. patients had a history of thoracic or abdominal surgery;
2. patients were IV to VI in the American Society of Anesthesiologists (ASA) physical status classification system;
3. patients had other malignancies;
4. patients had missing clinical data

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer undertaking resection by RAME were included. According to different perioperative management strategies, all eligible patients were divided into the ERAS group and conventional group.
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
time to first flatus | 2019-2022
  time to first flatus characterized by postoperative outcome
time to out-of-bed activity | 2019-2022
  time to out-of-bed activity characterized by postoperative outcome
time to liquid diet | 2019-2022
  time to liquid diet characterized by postoperative outcome
postoperative pain score | 2019-2022
  postoperative pain score characterized by postoperative outcome and was scored according to the numeric pain rating scale (NPRS) to assess the patient's pain on the first day after surgery.
duration of analgesic pump | 2019-2022
  duration of analgesic pump characterized by postoperative outcome
postoperative hospital stay | 2019-2022
  postoperative hospital stay characterized by postoperative outcome
ICU length of stay | 2019-2022
  ICU length of stay characterized by postoperative outcome
in-hospital mortality | 2019-2022
  in-hospital mortality characterized by postoperative outcome
incidence of various postoperative complications | 2019-2022
  incidence of various postoperative complications characterized by postoperative outcome

SECONDARY OUTCOMES:
postoperative chest drainage volume | 2019-2022
  postoperative chest drainage volume characterized by postoperative outcome
preoperative anesthesia time | 2019-2022
  preoperative anesthesia time characterized by intraoperative outcome
operation time | 2019-2022
  operation time characterized by intraoperative outcome
blood loss | 2019-2022
  blood loss characterized by intraoperative outcome
conversion rate | 2019-2022
  conversion rate characterized by intraoperative outcome
radicality of surgery | 2019-2022
  R0 resection was defined as > 1mm from all resection margins, R1 resection was defined as microscopic residual tumor, and R2 resection was defined as macroscopic residual tumor

CONTACTS AND LOCATIONS:
Overall Officials: Yidan Lin, MD, Study Director — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No